CLINICAL TRIAL: NCT00123318
Title: A Feasibility Study to Evaluate Adjuvant Chemoradiotherapy for Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: The Royal Australian and New Zealand College of Radiologists (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TROG 03.02
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Radiotherapy; Chemotherapy; Chemoradiation
MeSH Terms: conditions — Stomach Neoplasms | interventions — Epirubicin; Injections; Cisplatin; Fluorouracil; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Single-arm, non-randomised feasibility study to evaluate new regimen of adjuvant chemoradiotherapy (Epirubicin, Cisplatin, 5-Fluorouracil + radiotherapy)
  Interventions: Drug: epirubicin; Drug: cisplatin; Drug: 5-fluorouracil; Radiation: Radiotherapy

INTERVENTIONS:
Drug: epirubicin — 50mg/m2 IV day 1
  Other Names: Epirubicin Ebewe, Epirubicin Hydrochloride for Injection
Drug: cisplatin — 60mg/m2 IV day 1
  Other Names: Cisplatin Ebewe, Cisplatin Injection
Drug: 5-fluorouracil — 5-FU 200mg/m2/d IV 21 day continuous infusion Cont. infusional 5-FU 225mg/m2/day, 7 days/wk throughout entire period RT via CADD pump through PICC line
  Other Names: DBL Fluoruracil Injection BP, Efudix
Radiation: Radiotherapy — 45Gy 25 Fractions, 5 days/week for 5 weeks
  Other Names: Radiation

SUMMARY:
The purpose of this study is to determine the side-effects and effectiveness of a new type of chemoradiotherapy treatment for patients who have had surgery for stomach cancer. The treatment uses epirubicin, cisplatin, and 5-fluorouracil (ECF) chemotherapy together with radiotherapy.

DETAILED DESCRIPTION:
It has been shown recently in a study conducted in the USA (INT0116) that postoperative, adjuvant chemoradiotherapy improves survival for patients with gastric cancer. This treatment is relatively new and there remains debate regarding the optimal chemotherapy regimen and the optimal method of radiotherapy delivery. This study will evaluate a new regimen of adjuvant chemoradiotherapy for gastric cancer that employs ECF chemotherapy as the systemic component given before and after concurrent chemoradiation with continuous infusional 5-fluorouracil. Patients receive one cycle of ECF, followed 28 days later by chemoradiotherapy to a radiation dose of 45 Gy in 25 fractions over 5 weeks, and then one month later two further cycles of ECF are given. All patients are treated using multiple-field conformal radiation techniques.

The specific objectives of the study are:

* To detail the acute toxicity associated with this treatment.
* To determine the feasibility of the proposed concurrent chemoradiation regimen.
* To determine the feasibility of a standardized technique for radiation treatment planning and delivery.

The study will help to develop a common approach to the adjuvant treatment of gastric cancer, which is required before initiating further clinical trials in gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

All of the following must apply:

* Histologically proven adenocarcinoma of the stomach or gastro-oesophageal junction that is:

  1. completely resected with negative margins
  2. Stage T3,4 and/or N1,2 patients who have undergone a D2 nodal dissection can be entered on the study at the discretion of the treating clinician.
* Age greater than or equal to 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, 2
* Adequate organ function defined as follows:

  * Bone marrow: Haemoglobin greater than or equal to 90 g/L; Neutrophil count greater than or equal to 1.5 x 10^9 /L; Platelet count greater than or equal to 100 x 10^9 /L
  * Hepatic: Serum bilirubin less than or equal to 1.5 x ULN; AST and/or ALT less than or equal to 3.0 x ULN;
  * Renal: Serum creatinine less than or equal to 0.150 mmol/L, and calculated creatinine clearance greater than or equal to 50mL/min.
* Adequate oral nutrition (intake greater than or equal to 1500 calories/day). This is to be assessed by a dietician prior to commencing treatment.
* Disease which can be radically treated to 45 Gy with standard fractionation.
* Patient able to be treated with infusional 5-fluorouracil (5-FU) and ECF chemotherapy.
* Written informed consent

Exclusion Criteria:

None of the following must apply:

* Evidence of metastatic disease.
* Prior chemotherapy or radiotherapy
* Patients with other significant underlying medical conditions that may be aggravated by the study treatment or are not controlled.
* Pregnant or lactating females or female patients of childbearing potential who have not been surgically sterilized or are without adequate contraceptive measures.
* Cardiac failure (relevant to the use of epirubicin):

  * Patients with myocardial infarction within the last 6 months;
  * Patients with New York Heart Association class III/IV congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who develop grade 3 or grade 4 haematological and gastrointestinal acute toxicity | Final analysis will be at 3 years.
The percentage of patients who complete the planned chemoradiation protocol | Final analysis will be at 3 years.
The percentage of major radiotherapy protocol violations | Final analysis will be at 3 years.

SECONDARY OUTCOMES:
Median survival and overall survival at 3 years | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Leong, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (19):
- Australia (18):
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Nepean Cancer Care Centre, Penrith, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Mater QRI, Brisbane, Queensland
  - Royal Brisbane Hospital, Herston, Queensland
  - East Coast Cancer Centre, Tugun, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Launceston General Hospital, Launceston, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Andrew Love Cancer Care Centre, Geelong Hospital, Geelong, Victoria
  - Austin Health, Melbourne, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Hospital, Prahran, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- Christchurch Hospital, Christchurch, New Zealand

REFERENCES:
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au